CLINICAL TRIAL: NCT03942679
Title: Efficacy of Platelet Rich Plasma Injection in Comparison to Physical Therapy for Treatment of Chronic Partial Supraspinatus Tears
Brief Title: Platelet Rich Plasma and Supraspinatus Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS/17.08.79
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2019-05

CONDITIONS: Supraspinatus Tear
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRPinjection group (Other): Patients in this group will receive three ultrasound guided PRP injections in the supraspinatus tendon with one week interval (Ilhanli et al., 201
  Interventions: Other: PRP
- physiotherapy group (Other): Patients in this group will be treated with hot pack for 15 minutes, ultrasound in continuous mode (1.5 watt/cm2 for five minutes), trans-cutaneous electrical nerve stimulation in brief-intense mode for 15 minutes, range of motion (ROM), followed by stretching and strengthening exercises with 10 repeats 15 sessions (five sessions per week for three weeks
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: PRP — Patients in this group will receive three ultrasound guided PRP injections in the supraspinatus tendon with one week interval (Ilhanli et al., 2015). After the injection, patients will be instructed to limit the use of shoulder for at least 24 hours and to use cold therapy for pain. After the third injection, ROM, and stretching exercises will be allowed and one month after the end of injections, patients will be recommended to begin the strengthening program as tolerated. Exercise is performed with 10 repeats five sessions per week.
  Arms: PRPinjection group
Other: physiotherapy — Patients in this group will be treated with hot pack for 15 minutes, ultrasound in continuous mode (1.5 watt/cm2 for five minutes), trans-cutaneous electrical nerve stimulation in brief-intense mode for 15 minutes, range of motion (ROM), followed by stretching and strengthening exercises with 10 repeats 15 sessions (five sessions per week for three weeks). After the physical therapy, the exercise program will be continued as homework during the follow-up period.
  Arms: physiotherapy group

SUMMARY:
Rheumatology and Rehabilitation Department, Mansoura University Hospital. Forty patients with chronic partial supraspinatus tears will be included in the study. The diagnosis of the supraspinatus tear will be made by ultrasound examination

DETAILED DESCRIPTION:
At inclusion in the study, demographic data (age, gender, duration of complaints, and body mass index) will be recorded.

Randomization

Patients will be randomized into two matched groups:

A) PRP-Injection Group - Patients in this group will receive three ultrasound guided PRP injections in the supraspinatus tendon with one week interval (Ilhanli et al., 2015). After the injection, patients will be instructed to limit the use of shoulder for at least 24 hours and to use cold therapy for pain. After the third injection, ROM, and stretching exercises will be allowed and one month after the end of injections, patients will be recommended to begin the strengthening program as tolerated. Exercise is performed with 10 repeats five sessions per week.

B) Physical Therapy Group - Patients in this group will be treated with hot pack for 15 minutes, ultrasound in continuous mode (1.5 watt/cm2 for five minutes), trans-cutaneous electrical nerve stimulation in brief-intense mode for 15 minutes, range of motion (ROM), followed by stretching and strengthening exercises with 10 repeats 15 sessions (five sessions per week for three weeks). After the physical therapy, the exercise program will be continued as homework during the follow-up period.

Patients in t

ELIGIBILITY:
Inclusion Criteria:

chronic partial supraspinatus tears will be included in the study

Exclusion Criteria:

age > 80 years, pregnancy, full thickness supraspinatus tears, other rotator cuff lesions with/without supraspinatus tears, systemic disorders such as diabetes rheumatoid arthritis, hematological diseases (co-agulopathy),

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
change of pain from base line | immediately before injection,6 weeks after injection,12 weeks after injection
  The VAS-pain score is composed of a continuous horizontal line. This line is 100 mm in length. To measure the intensity of pain, the score is anchored by (0 score = no pain) at one end and (100 score = worst imaginable pain) on the other end. The patient places a mark to the VAS line at the point which represents the intensity of his pain
change of range of motion from base line | immediately before injection,6 weeks after injection,12 weeks after injection
  III. Examination of passive and active range of motion using goniometer based on the description of norkin and white as following
  * Abduction ;170
  * Adduction :50
  * Flexion :165
  * Extension:60
  * Internal rotation at 90 abduction :70
  * External rotation at 90 abduction :100

SECONDARY OUTCOMES:
change of shoulder index score from base line | immediately before injection,6 weeks after injection,12 weeks after injection
  •Disability and health related quality of life will be measured using DASH shoulder rating scale.
change of ultrasound pathology from base line | immediately before injection,,12 weeks after injection
  •US documented pathology will be assessed at diagnosis and at 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Magdy Shaat, Al Mansurah, Dakahlia Provence, Egypt

IPD SHARING:
Plan to Share IPD: Undecided